CLINICAL TRIAL: NCT07362498
Title: Spatiotemporal Dynamics of Antimalarial Drug Resistance in Western Kenya During a Pilot Multiple First-line Treatment for Uncomplicated Malaria Study: Molecular Evidence of Resistance Saturation and Emerging Artemisinin Tolerance
Brief Title: Health Systems Implementation and Molecular Surveillance of Multiple First-Line Treatments for Uncomplicated Malaria in Western Kenya
Status: Completed | Type: Observational
Sponsor: Strathmore University (Other)
Collaborators: Medicines for Malaria Venture (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); Kenya Ministry of Health (Other Government); National Malaria Control Programme, Kenya (Unknown); Homa Bay County Government, Kenya (Unknown); Migori County Government, Kenya (Unknown); Kenya Medical Supplies Authority (KEMSA), Kenya (Unknown)
Responsible Party: Principal Investigator, Andrew Cole, Research Scientist, Strathmore University
Other Study IDs: SU-MFT-2020-001; PO20/00538 (Other Grant/Funding Number: Medicines for Malaria Venture (MMV))
Record Dates: First submitted 2026-01-01; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Malaria Falciparum
Keywords: malaria; Drug Resistance; Multiple first-line therapies; Plasmodium falciparum; Molecular surveillance
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — This observational molecular surveillance study was non-randomized. Multiple first-line therapies (MFTs) were deployed by health authorities as a health systems implementation program (Reference 34). The research team conducted observational molecular analysis only and did not assign treatments.
  Homa Bay Mainland received 8-month ACT cycling: AL baseline, then DHA-PIP, AS+AQ, and return to AL. Mfangano Island received extended 39-month AS+PYD deployment. Migori County continued AL monotherapy throughout (control).
  Dried blood spots (DBS) were collected from malaria-positive, de-identified laboratory samples at four time-points: T1 (Sep 2020, AL all sites), T2 (Aug-Oct 2021, DHA+PIP Homa Bay Mainland, AS+PYD 12 months Mfangano), T3 (May-Jul 2022, AS+AQ Homa Bay, AS+PYD Mfangano), T4 (Nov 2023-Jan 2024, Mfangano extended follow-up). Samples were analyzed by targeted amplicon deep sequencing for antimalarial resistance markers in dhfr, dhps, mdr1, and k13 genes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Homa Bay Mainland: MFT Adaptive Cycling: Sequential deployment of multiple first-line artemisinin-based combination therapies using 8-month adaptive cycling with crowding-out approach. Treatment sequence: Baseline artemether-lumefantrine (AL) followed by dihydroartemisinin-piperaquine (DHA-PIP) for 8 months, then artesunate-amodiaquine (AS+AQ) for 8 months, then return to AL for 8 months. Approximately 40,000 patients treated across multiple health facilities. Note: This observational molecular surveillance study analyzed resistance markers from samples collected during MFT deployment by health authorities (described in Reference 34). Arms represent different drug deployment contexts in which molecular surveillance was conducted. No intervention by research team; observational analysis only.
  Interventions: Drug: Artemether + Lumefantrine; Drug: Dihydroartemisin-piperaquine; Drug: Artesunate-Amodiaquine (AS-AQ)
- Mfangano Island: MFT Extended Deployment: Extended deployment of a single alternative artemisinin-based combination therapy in a geographically isolated island setting. Treatment sequence: Baseline artemether-lumefantrine (AL) followed by pyronaridine-artesunate (AS+PYD) for extended 39-month period. Approximately 21,000 patients treated. This arm assessed health systems feasibility and molecular resistance dynamics with prolonged single MFT deployment in a relatively closed transmission environment since minimal data was available owing to AS+PYD recency of formulary inclusion. Note: This observational molecular surveillance study analyzed resistance markers from samples collected during MFT deployment by health authorities (described in Reference 34). Arms represent different drug deployment contexts in which molecular surveillance was conducted. No intervention by research team; observational analysis only.
  Interventions: Drug: Artemether + Lumefantrine; Drug: Pyronaridine - artesunate
- Migori: Control: Continued artemether-lumefantrine (AL) as the only ACT throughout the entire study period as per Kenya national malaria treatment guidelines. Served as comparison group for health systems outcomes and molecular resistance surveillance. Approximately 32,835 patients treated. This arm represents standard of care without MFT intervention. Note: This observational molecular surveillance study analyzed resistance markers from samples collected during MFT deployment by health authorities (described in Reference 34). Arms represent different drug deployment contexts in which molecular surveillance was conducted. No intervention by research team; observational analysis only.
  Interventions: Drug: Artemether + Lumefantrine

INTERVENTIONS:
Drug: Artemether + Lumefantrine — Fixed-dose artemisinin-based combination therapy containing artemether and lumefantrine with dosage calculated by weight-bands according to manufacturers recommendations. Administered orally twice daily for 3 days (6 doses total). Used as baseline treatment across all study arms and continued throughout study period in comparison county. First-line treatment for uncomplicated malaria in Kenya. Supplied by Kenya Medical Supplies Authority through routine government procurement.
Drug: Dihydroartemisin-piperaquine — Fixed-dose artemisinin-based combination therapy containing dihydroartemisinin and piperaquine with dosage calculated by weight-bands according to manufacturers recommendations. Administered orally once daily for 3 days (3 doses total). Deployed in Homa Bay Mainland for 8 months during adaptive cycling. Donated by Tridem Pharma Ltd through Tridem Pharma Kenya. WHO-recommended ACT for uncomplicated falciparum malaria.
  Groups: Homa Bay Mainland: MFT Adaptive Cycling
Drug: Artesunate-Amodiaquine (AS-AQ) — Fixed-dose artemisinin-based combination therapy. Administered orally once daily for 3 days (3 doses total) with dosage calculated by weighted-bands according to manufacturers recommendations. Deployed in Homa Bay Mainland for 8 months during adaptive cycling following DHA-PIP deployment. Donated by Sanofi through Surgi Pharm Ltd Kenya. WHO-recommended ACT for uncomplicated falciparum malaria.
  Groups: Homa Bay Mainland: MFT Adaptive Cycling
Drug: Pyronaridine - artesunate — Fixed-dose artemisinin-based combination therapy containing pyronaridine and artesunate (granule formulation) with dosage calculated by weighted-bands according to manufacturers recommendations. Administered orally once daily for 3 days (3 doses total). Deployed in Mfangano Island for extended 39-month period. Donated by Shin Poong Pharmaceuticals Co. Ltd, Republic of South Korea. WHO-recommended ACT for uncomplicated falciparum malaria, registered in Kenya but not yet included in national treatment guidelines at time of study hence the need for an extended observational follow-up period.
  Groups: Mfangano Island: MFT Extended Deployment

SUMMARY:
This implementation study evaluated the health systems feasibility, economic costs, and stakeholder acceptability of deploying multiple first-line therapies (MFTs) that were of the artemisinin-based combination therapies (ACTs) type, for uncomplicated malaria in Western Kenya. The study included a nested observational molecular surveillance of antimalarial resistance markers in Plasmodium falciparum parasites. The implementation program involved adaptive cycling of four ACTs across 28 health facilities over 28 months (June 2020 - October 2022) with and extension to January 2024 in one geographic area (Mfangano Island). Health systems outcomes (feasibility, costs, acceptability) are reported in Cole et al., Malaria Journal 2024. Molecular surveillance outcomes (resistance marker prevalence and temporal trends) are reported in a companion manuscript currently under peer-review.

DETAILED DESCRIPTION:
BACKGROUND: Artemisinin-based combination therapies (ACTs) are first-line treatment for uncomplicated malaria in sub-Saharan Africa, but emerging artemisinin partial resistance threatens efficacy. Multiple first-line treatments (MFTs) represent a proposed strategy to delay resistance emergence by deploying several ACTs simultaneously, sequentially, or using other strategies rather than relying on a single first-line therapy.

STUDY DESIGN: This 28-month implementation program (June 2020 - October 2022) with and extension only on Mfangano Island until January 2024, deployed adaptive cycling of four artemisinin-based combinations across health facilities in Western Kenya using geographic allocation:

INTERVENTION COUNTY - HOMA BAY:

* Homa Bay Mainland (n=approximately 40,000 patients treated): Sequential deployment with 8-month cycling using crowding-out approach: Baseline (AL) → DHA-PIP (8 months) → AS+AQ (8 months) → AL (8 months)
* Mfangano Island (n=approximately 21,000 patients treated): Extended single MFT deployment: Baseline (AL) → AS+PYD (39 months). This extension allowed longer follow-up surveillance of the most recent combination ACT in Kenya where data was not previously monitored.

COMPARISON COUNTY - MIGORI:

- Continued artemether-lumefantrine (AL) monotherapy throughout study period (n=32,835 patients treated) PARTICIPANTS: Adults and children ≥5 years diagnosed with uncomplicated Plasmodium falciparum malaria at participating health facilities. Excluded: pregnant women and children <5 years due to medication restrictions and lack of pediatric formulations.

OUTCOMES MEASURED:

Primary Outcomes (reported in Cole et al., Malaria Journal 2024):

1. Health systems feasibility was assessed through commodity management, human resources adequacy, information system functionality, and implementation barriers/facilitators analysis
2. Economic costs of MFT deployment including start-up and implementation phases, calculated per facility and per patient were sought after
3. Stakeholder acceptability among policymakers, healthcare workers, and patients assessed through key informant interviews and surveys was analyzed.

Secondary Outcomes (reported in companion manuscript recently submitted for peer-review):

1. Prevalence of antimalarial resistance markers in dhfr (N51I, C59R, S108N, I164L), dhps (S436H, A437G, K540E, A581G), mdr1 (N86Y, Y184F), and k13 (A578S, A675V) genes
2. Temporal trends in resistance marker prevalence over four timepoints (September 2020, August-October 2021, May-July 2022, November 2023-January 2024)
3. Geographic distribution of resistance patterns across study sites
4. Complexity of infection (COI) determined by molecular methods

METHODS:

* Sample collection: Dried blood spots (n=310) from malaria-positive patients at four timepoints
* Molecular analysis: Targeted amplicon deep sequencing using Oxford Nanopore Technology
* Health systems assessment: Semi-structured questionnaires, key informant interviews, exit interviews, cost analysis using activity-based costing
* Statistical analysis: Chi-square tests, Cochran-Armitage trend tests, machine learning models for resistance prediction SETTING: Government and faith-based health facilities in Homa Bay County facilities received MFTs and Migori County (control) where AL was the only ACT used in Western Kenya, a malaria-endemic region with high transmission intensity.

ETHICAL APPROVAL: Strathmore University Institutional Scientific and Ethics Review Committee (SU-ISERC 1730/20) and Kenya National Commission for Science, Technology and Innovation (NACOSTI).

ELIGIBILITY:
Inclusion Criteria:

* Age 5 years or older
* Clinical diagnosis of uncomplicated malaria
* Confirmed Plasmodium falciparum infection by rapid diagnostic test (RDT) or microscopy
* Presenting at participating health facility for malaria treatment
* Able and willing to provide informed consent (or parental/guardian consent for minors under 18 years)
* Resident of study catchment area
* For molecular surveillance substudy: willingness to provide dried blood spot sample

Exclusion Criteria:

* Pregnant women (due to contraindications for some study medications in first trimester and lack of safety data)
* Children under 5 years of age (due to lack of pediatric formulations for some study medications)
* Severe or complicated malaria requiring parenteral treatment or hospitalization
* Known hypersensitivity or contraindication to any of the study artemisinin-based combination therapies
* Unable to take oral medications
* Previous participation in current treatment episode (repeat visits)
* Concurrent participation in other interventional malaria treatment studies

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with uncomplicated Plasmodium falciparum malaria at participating government and faith-based health facilities in Homa Bay County and Migori County, Western Kenya, a malaria-endemic region with high transmission intensity.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Health Systems Feasibility - Commodity Management Score | June 2020 to January 2024
  Assessment of drug supply chain functionality including quantification accuracy, stock management, and distribution logistics. Measured using structured health facility assessment checklist scoring five domains: (1) drug availability, (2) stock-out frequency, (3) quantification accuracy, (4) storage conditions, (5) distribution timeliness. Score range 0-100 where higher scores indicate better commodity management. Assessed at 28 health facilities.
Health Systems Feasibility - Human Resources and Information Systems Score | June 2020 to January 2024
  Assessment of human resources adequacy and health information system functionality. Measured using structured facility assessment scoring: (1) healthcare worker availability, (2) training completion rates, (3) reporting tool adoption, (4) KHIS2 system functionality. Score range 0-100 where higher scores indicate better health systems capacity. Assessed at 28 health facilities.
Stakeholder Acceptability - Composite Acceptability Score | June 2020 - January 2024
  Composite measure of MFT deployment acceptability among three stakeholder groups: policymakers, healthcare workers, and patients. Measured through: (1) key informant interviews (n=85) using semi-structured guides rated on 5-point Likert scale, (2) patient exit interviews assessing treatment satisfaction (5-point scale), (3) healthcare worker surveys assessing implementation feasibility (5-point scale). Composite score calculated as mean across all stakeholder groups. Range 1-5 where higher scores indicate greater acceptability.
Economic Costs of Multiple First-Line Treatment Implementation | June 2020 to January 2024
  Total economic costs of MFT deployment calculated using activity-based costing approach with ingredient method. Includes start-up phase costs (training, IEC materials, reporting tool revision, KHIS2 updates, sensitization) and implementation phase costs (drug procurement, distribution, refresher training, quantification). Costs tracked prospectively from documents, receipts, and market prices. Reported as: (1) total economic vs financial costs in USD, (2) costs by category, (3) costs by funding source, (4) unit cost per facility covered in USD, (5) unit cost per patient treated in USD. Start-up costs annualized over 3-year useful life at 3% discount rate.

SECONDARY OUTCOMES:
Prevalence of Antimalarial Resistance Markers | September 2020 to January 2024
  Frequency of known resistance-associated mutations measured as percentage allele frequency (%) for all markers.
  Assessed in four Plasmodium falciparum genes: (1) dhfr - dihydrofolate reductase (codons N51I, C59R, S108N, I164L), (2) dhps - dihydropteroate synthase (codons S436H, A437G, K540E, A581G), (3) mdr1 - multidrug resistance protein 1 (codons N86Y, Y184F), and (4) k13 - kelch13 propeller domain (codons A578S, A675V).
  Determined by targeted amplicon deep sequencing of dried blood spots (n=310) using Oxford Nanopore Technology. Allele frequencies calculated as percentage of reads supporting each allele (range 0-100%). Infections classified as wild-type, mutant, or mixed. Haplotype frequencies determined from microhaplotype analysis.
Change in Antimalarial Resistance Marker Prevalence Over Time (Cochran-Armitage Trend Test) | Four time-points over 40 months: T1 (September 2020), T2 (August - October 2021), T3 (May - July 2022), T4 (November 2023 - January 2024)
  Change in resistance marker prevalence measured as percentage point difference between timepoints, with statistical significance assessed using Cochran-Armitage test for trend.
  Measured over four serial cross-sectional timepoints: T1 (September 2020, baseline when AL used at all sites), T2 (August-October 2021, during MFT deployment), T3 (May-July 2022, continued MFT deployment), T4 (November 2023-January 2024, extended follow-up Mfangano Island only).
  Primary measurement: percentage point change in allele frequency from T1 to T3 (all sites, n=240 balanced comparison). Secondary measurement: percentage point change T1 to T4 (Mfangano Island only, n=111 extended surveillance). Statistical significance determined using Cochran-Armitage test for trend (P<0.05 significant). Assessed separately for each individual mutation and for combined haplotypes.
Geographic Distribution of Antimalarial Resistance Markers | September 2020 - January 2024
  Comparison of resistance marker prevalence across three geographic study areas: (1) Homa Bay Mainland (intervention with 8-month adaptive cycling), (2) Mfangano Island (intervention with extended single MFT), and (3) Migori County (comparison with continued AL single ACT use). Statistical comparisons using chi-square tests for categorical variables and Fisher's exact tests for intervention vs comparison effects. Analysis accounts for unbalanced sampling design with extended follow-up only for Mfangano Island.
Complexity of Infection in Plasmodium falciparum | September 2020 - January 2024
  Mean complexity of infection (COI) defined as the number of genetically distinct parasite clones per infection. Determined using two complementary methods: (1) ama1 genotyping counting maximum number of distinct alleles at polymorphic positions (n=310 samples), and (2) direct haplotype counting from targeted amplicon deep sequencing reads (n=176 samples with sufficient coverage). Infections classified as monoclonal (COI=1) or polyclonal (COI>1). Geographic variation assessed using Kruskal-Wallis test with post-hoc Dunn's test. Results provide context for interpretation of resistance marker data in high-transmission setting.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Kokwaro, PhD, FKNAS, FAAS, Study Director — Institute of Healthcare Management, Strathmore University
Locations (2):
- Kenya (2):
  - Homa Bay County Health Facilities, Homa Bay, Homa Bay County
  - Migori County Teaching and Referral Hospital, Migori, Migori County Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole A, Chege T, Aman R, Githuka G, Muga R, Aspinall A, Kokwaro G. Health system challenges and facilitators associated with adaptive cycling deployment of multiple first-line treatment for uncomplicated malaria: a pilot study in a malaria-endemic region of Kenya. Malar J. 2025 Oct 10;24(1):328. doi: 10.1186/s12936-025-05580-7. PMID 41074071
- See also: Published health systems outcomes from parent implementation study — https://doi.org/10.1186/s12936-025-05580-7